CLINICAL TRIAL: NCT04480632
Title: Therapeutic Plasmapheresis in Critically Ill Adult Patients With COVID-19 Confirmed Diagnosis / Plasmaféresis terapéutica en Pacientes Adultos críticamente Enfermos Con diagnóstico Confirmado de COVID-19
Brief Title: Therapeutic Plasmapheresis in Critically Ill Adult Patients With COVID-19 Confirmed Diagnosis
Acronym: PLASMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2020-01200
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; Convalescent plasma; Intensive Care Unit; Critical illness
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Intervention Model Description: Quasi-experimental and open-label intervention study. In this study, the application of convalescent plasma is considered as an intervention, but randomization will not be performed by investigators; one arm will be patients who received ABO compatible convalescent plasma and the comparison group will be those patients with intervention indication but without compatible ABO plasma units within the institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABO compatible convalescent plasma (Experimental): A 500 ml dose of convalescent plasma (from a single donor or two 250 ml units from one or two donations) collected by apheresis will be administered. In case of plasma storage, plasma unit will be thawed following parameters of blood bank. Administration will take place slowly and over the course of four hours. When two 250 ml units are administered, second unit must be administered after the first unit in a period not exceeding 12 hours.
  Interventions: Biological: Convalescent plasma
- Usual care (No Intervention): Usual medical care for critically ill patients at ICU

INTERVENTIONS:
Biological: Convalescent plasma — ABO compatible convalescent plasma obtained from from recovered COVID-19 patients
  Arms: ABO compatible convalescent plasma

SUMMARY:
Introduction: The SARS-CoV-2 outbreak has left more than two million infected worldwide in the first four months of COVID-19 epidemic. To date, there is no specific treatment for the disease and in critically ill patients there is an additional challenge in controlling the systemic inflammatory response, which is characterized by cytokine storm, alteration in coagulation and endothelial activation in addition to infection. Strategies used in previous viral epidemics, such as convalescent plasma, are therapeutic options to rescue, especially in individuals with a critical presentation of the disease.

Aim: To establish clinical response of critically ill patients with COVID-19 who received convalescent plasma from subjects recovered from SARS-CoV-2 during their stay in Intensive Care Unit at Fundación Cardiovascular de Colombia (Hospital Internacional de Colombia).

Methodology: Quasi-experimental study (no randomization will be performed). Adult patients who meet selection criteria will receive 500 ml of ABO compatible convalescent plasma, obtained by apheresis from patients recovered from SARS-CoV-2 infection. The main outcome will be in-hospital mortality at 30 days, while indication for ventilatory support (intubation) and adverse events at thirty days will be evaluated as secondary outcomes, compared to subjects receiving usual treatment for clinical sign and symptoms given the absence of ABO compatible plasma units. A survival analysis will be performed using Kaplan-Meier method and association strength will be reported using HR and 95% CI crude and adjusted for confounding variables.

Expected results: It is expected to know the clinical and paraclinical response of patients receiving convalescent plasma in our institution, as well as to establish their probability of survival and its associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Over 18 years old
* Patients with confirmed infection by COVID-19 (positive real-time PCR) in ICU with:
* Respiratory failure receiving ventilatory support and high parameters
* Severe pneumonia with rapid progression
* Ability to sign informed consent

Exclusion Criteria:

* Pregnant women
* Contraindication of plasma administration due to history of anaphylaxis during transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  In-hospital mortality after administration of ABO compatible convalescent plasma or indication (but not plasmapheresis for absence of compatible convalescent plasma) for comparison group

SECONDARY OUTCOMES:
Incidence of renal replacement therapy | 30 days
  Number of patients with medical indication of hemodialysis or peritoneal dialysis for acute renal failure
Incidece of adverse events | During tranfusion until 24 hours after.
  Number of patients with Alergic reaction, Anaphylaxis, Severe thrombotic events, Transfusion-related acute lung injury (TRALI)], Transfusion-associated circulatory overload (TACO)], Antibody-Dependent Enhancement (ADE)]

CONTACTS AND LOCATIONS:
Overall Officials: Norma Serrano, MD, Principal Investigator — Research, development and innovation director
Locations (1):
- Hospital Internacional de Colombia, Piedecuesta, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Hui DS. Severe acute respiratory syndrome (SARS): lessons learnt in Hong Kong. J Thorac Dis. 2013 Aug;5 Suppl 2(Suppl 2):S122-6. doi: 10.3978/j.issn.2072-1439.2013.06.18. PMID 23977432
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Keith P, Day M, Perkins L, Moyer L, Hewitt K, Wells A. A novel treatment approach to the novel coronavirus: an argument for the use of therapeutic plasma exchange for fulminant COVID-19. Crit Care. 2020 Apr 2;24(1):128. doi: 10.1186/s13054-020-2836-4. No abstract available. PMID 32241301
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Ahn JY, Sohn Y, Lee SH, Cho Y, Hyun JH, Baek YJ, Jeong SJ, Kim JH, Ku NS, Yeom JS, Roh J, Ahn MY, Chin BS, Kim YS, Lee H, Yong D, Kim HO, Kim S, Choi JY. Use of Convalescent Plasma Therapy in Two COVID-19 Patients with Acute Respiratory Distress Syndrome in Korea. J Korean Med Sci. 2020 Apr 13;35(14):e149. doi: 10.3346/jkms.2020.35.e149. PMID 32281317